CLINICAL TRIAL: NCT00245817
Title: Coronary Artery Bypass Grafting (CABG) Patients in the Rehabilitation Phase. A Randomised Controlled Trial.
Brief Title: HINCAB-study. Home Based Intervention in Nursing for Coronary Artery Bypass Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Responsible Party: Principal investigator: Irene Lie, PhD student, Ullevaal University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: HINCAB
Record Dates: First submitted 2005-10-27; First posted 2005-10-28 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2010-12

CONDITIONS: Anxiety; Depression
Keywords: Anxiety. Depression. HRQOL. Psycho-educative intervention
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: HINCAB — Psycho-educative intervention performed 2 and 4 weeks after surgery

SUMMARY:
HINCAB-study is a single senter, prospective, randomised controlled trial. The aim of the study is to test the effect of a home based intervention program. The hypothesis of the study is that a home based intervention will influencing coping strategies in the CABG-patients rehabilitation phase, reduce symptoms and improve health related quality of life.

DETAILED DESCRIPTION:
Research has shown better quality of life for patients after CABG. At the same point of time studies shows that patients experience anxiety and depression years after surgery. Anxiety and depression appear frequently at the same time and strengthen each other. Studies underline that CABG-patients especially the first month after surgery want follow-up by health care provider. Anxiety and depression are assessed as independent risk factors for morbidity and death in heart patients.

203 CABG-patients were randomised into the study. Both patient group, the experimental- and control group, answered the same three standardised questionnaires before surgery, 6 weeks and 6 months after surgery. The questionnaires are Hospital Anxiety and Depression Scale (HADS), Seattle Angina Questionnaire (SAQ) and SF-36.

The intervention consist of two home visits 2 and 4 weeks after CABG undertaken by project leader. The intervention protocol has been approved by The Norwegian Committee for Medical Research Ethics.

Knowledge from this study may generate a basis for clinical guidelines and patient pathways. Results from this study will show if the home based intervention in the future will be performed for only a risk group of about 20 % that have responded best to the intervention. In the future the intervention also may be individualized electronically.

ELIGIBILITY:
Inclusion Criteria: Elective CABG-patients admitted to Ullevål University Hospital. The patients must be capable, physical and mental to fill in all questionnaires. In addition, to be capable to read and understand Norwegian. Driving distance maximum three hours each way.

Exclusion Criteria: Patients with combined surgery (coronary- and valve replacement surgery). Emergency surgery. Redo. Patients that related to surgery experience cerebral insult, mediastinitis or become intensive care patients will be excluded from this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2003-08; Primary Completion 2005-01 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Anxiety and depression symptoms | 6 months

SECONDARY OUTCOMES:
Health related quality of life | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Irene Lie, PhD student, Principal Investigator — Ullevaal University Hospital; Eli H Bunch, Professor, Study Chair — Institute of Nursing and Health Science
Locations (1):
- Ullevål University Hospital, Oslo, Norway

REFERENCES:
- [Result] Lie I, Arnesen H, Sandvik L, Hamilton G, Bunch EH. Health-related quality of life after coronary artery bypass grafting. The impact of a randomised controlled home-based intervention program. Qual Life Res. 2009 Mar;18(2):201-7. doi: 10.1007/s11136-008-9438-y. Epub 2009 Jan 25. PMID 19169899
- [Result] Lie I, Arnesen H, Sandvik L, Hamilton G, Bunch EH. Effects of a home-based intervention program on anxiety and depression 6 months after coronary artery bypass grafting: a randomized controlled trial. J Psychosom Res. 2007 Apr;62(4):411-8. doi: 10.1016/j.jpsychores.2006.11.010. PMID 17383492
- [Result] Lie I, Arnesen H, Sandvik L, Hamilton G, Bunch EH. Predictors for physical and mental health 6 months after coronary artery bypass grafting: a cohort study. Eur J Cardiovasc Nurs. 2010 Dec;9(4):238-43. doi: 10.1016/j.ejcnurse.2010.02.001. Epub 2010 Mar 9. PMID 20219433
- [Result] Lie I, Bunch EH, Smeby NA, Arnesen H, Hamilton G. Patients' experiences with symptoms and needs in the early rehabilitation phase after coronary artery bypass grafting. Eur J Cardiovasc Nurs. 2012 Mar;11(1):14-24. doi: 10.1016/j.ejcnurse.2010.09.004. PMID 21030311